CLINICAL TRIAL: NCT02306356
Title: Internet-delivered Treatment for Children With Anxiety Disorders in a Rural Area; an Open Trial in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: BUP Östersund (Unknown)
Responsible Party: Principal Investigator, Eva Serlachius, associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1225-31/4
Record Dates: First submitted 2014-09-27; First posted 2014-12-03 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Specific Phobia; Separation Anxiety; Generalized Anxiety Disorder
MeSH Terms: conditions — Phobia, Specific; Anxiety, Separation; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional (Experimental): Behavioral: Internet-delivered Cognitive Behavior Therapy
  Interventions: Behavioral: Internet-delivered Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavior Therapy

SUMMARY:
An open trial will be conducted at the Child and Mental Health Service (CAMHS) unit in the rural county Jämtland in Sweden to test the feasibility and efficacy of Internet-delivered Cognitive Behavior Therapy (ICBT) for children with anxiety disorders in a clinical setting. 20 children with a principal diagnosis of Generalized Anxiety Disorder (GAD), separation anxiety, specific phobia and their parents will be recruited from the CAMHS-center in Östersund. They will receive 12 weeks of therapist-supported ICBT and will be assessed by clinician ratings and child- and parent-reports at baseline, post-treatment and 3 month follow-up. The primary outcome measures the Clinical Global Impressions - Severity scale (CGI-S). Secondary outcome measures include clinician rated global functioning, and child and parent-rated anxiety and functioning.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 years of age
* Fulfilling diagnostic criteria for Generalized Anxiety Disorder (GAD), Separation anxiety, Specific phobia
* Ability to read and write Swedish
* Daily access to the internet
* A parent that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 3 months prior to baseline assessment

Exclusion Criteria:

* Diagnosed autism spectrum disorder or Attention-deficit/hyperactivity disorder (ADHD), or principal primary disorder other than GAD, Separation anxiety, Specific phobia
* Acute/severe psychiatric problems such as suicidal risk or severe depression
* Ongoing psychological treatment for anxiety disorders
* Ongoing child custody dispute or abuse in the family

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impressions - severity (CGI-S) | baseline, post-treatment (12 weeks), follow-up (3 months)
  Change in CGI-s from baseline to post-treatment and follow-up

SECONDARY OUTCOMES:
Children´s Global Assessment Scale (CGAS | Baseline, post-treatment (12 weeks), follow-up (3 months)
Spence Child Anxiety Scale C/P (SCAS-C/P) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Penn State Worry Questionnaire (PSWQ) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Separation Anxiety Index (SAI) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Fear Survey Schedule for Children - Revised (FSSC-R) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Child Sheehan Disability Scale (CSDS) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Child Depression Inventory (CDI) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Hospital Anxiety Depression Scale (HAD) | Baseline, post-treatment (12 weeks), follow-up (3 months)
Client Satisfaction Scale (CSS) | post-treatment (12 weeks)
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post-treatment (12 weeks), follow-up (3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Mental Health Services Östersund, Östersund, Jämtland County, Sweden